CLINICAL TRIAL: NCT01258335
Title: Short Term Ocular Safety Assessment of High Dose Omega-3 Supplementation for Age-Related Macular Degeneration.
Brief Title: Omega-3-fatty Acids on Age-related Macular
Acronym: Omega 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid Atlantic Retina (Other)
Collaborators: LifeGuard (Unknown)
Responsible Party: Dr. Allen Ho, Principal Investigator, Mid Atlantic Retina
Allocation: Randomized | Masking: Triple | Purpose: Prevention
Other Study IDs: 08-887
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Aged Macular Degeneration
MeSH Terms: interventions — Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega 3 Fatty acids (Active Comparator): II. Study arms:
  a. Participants in the dry AMD study group will be randomized into two arms with a 4:1 ratio: i. Omega-3-fatty acids 4 gm oral daily (Total:840mg EPA/2520mg DHA) (1:3 ratio of EPA to DHA) ( 6 capsules fatty acids)
  Interventions: Dietary Supplement: Omega 3
- Olive Oil (Placebo Comparator): ii. Placebo oral daily (6 softgel capsules, each contains 1100 mg olive oil)
  Interventions: Other: Olive Oil

INTERVENTIONS:
Dietary Supplement: Omega 3 — Omega-3-fatty acids 4 gm oral daily (Total:840mg EPA/2520mg DHA) (1:3 ratio of EPA to DHA) ( 6 capsules fatty acids)
  Arms: Omega 3 Fatty acids
Other: Olive Oil — ii. Placebo oral daily (6 softgel capsules, each contains 1100 mg olive oil)
  Arms: Olive Oil

SUMMARY:
Aim: To demonstrate the short-term multi focal electroretinogram (mfERG) effect of oral omega-3-fatty acids in the triglyceride form on dry age-related macular degeneration (AMD).

Null hypothesis: Omega-3-fatty acids do not affect the mfERGs of patients with dry AMD.

DETAILED DESCRIPTION:
There is a growing amount of basic science data supporting the use of omega 3 fatty acids in AMD. Koto et al. report that eicosapentaenoic acid, a major omega-3 polyunsaturated fatty acid, prevents CNVM in mice. Conner et al. report in Nature Medicine that increased dietary intake of omega-3-polyunsaturated fatty acids reduces pathological retinal angiogenesis in mice. Miyauchi et al. looked at ERG outcomes in rabbits. They report that an intraperitoneal injection of docosahexaenoic acid given 5 hours before IOP induced ischemia resulted in better ERG amplitudes than controls. Docosahexaenoic acid appears to protect against transient retinal ischemia.

Clinical data on this topic is scarce. A systemic review was published in Retina in 2007 (Hodge, et al.) outlining the limited data. A recent meta-analysis by Chong et al. of nine studies found a high dietary intake of omega-3 fatty acids decreased risk of late AMD by 38%, though the current literature is insufficient to support routine consumption to prevent AMD. Scorolli et al. conducted a randomized control trial on 35 bilateral wet AMD patients receiving photodynamic therapy with our without vitamin E, linolenic acid, alpha-linolenic acid, and docosahexaenoic acid (DHA). The latter two are omega-3-fatty acids. Patients in the polyunsaturated fatty acid (PUFA) group had significantly shorter recovery time after macular flash. Visually acuity was not statistically different between the two groups. Feher et al. conducted a randomized control trial using acetyl-L-carnitine, omega-3 fatty acids, and coenzyme Q10 (Phototrop). They report findings that strongly suggest that an appropriate combination of compounds that affect mitochondrial lipid metabolism may improve and subsequently stabilize visual functions, and it may also improve fundus alterations in patients affected by early AMD. The Blue Mountain Eye Study, a cohort study, reports a regular diet high in omega-3 polyunsaturated fat, especially from fish, seems to protect against early and late ARM. Seddon et al. performed a clinic-based case-control study across five centers, concluding diets high in omega-3 fatty acids and fish are inversely associated with risk for AMD when intake of linoleic acid was low. Augood et al. published a cross-sectional study of 105 cases, reporting eating oily fish at least once per week compared with less than once per week decreased the odds ratio for neovascular AMD by half.

Few authors have evaluated the role of ERG in treating AMD. A recent review by Gerth concludes ERG is an important tool in assessing retinal function in AMD and as an outcome measure. Multifocal ERG, possibly combined with other tests, has the greatest value. Hishihara et al. have evaluated the amplitude and implicit time changes in neovascular AMD using focal macular ERGs.

ELIGIBILITY:
Inclusion Criteria:

i. >49 year old women and men for the dry AMD arms. >20 year old for the normal retina arm.

1. No specific race/ethnic background requirements

Exclusion Criteria:

i. For dry AMD groups, all patients will be included, regardless of prior or concomitant treatment, and regardless of stage of disease.

ii. Patients already taking omega-3-fatty acids will be excluded. iii. Women of childbearing age with positive urine pregnancy tests or with plans to conceive during the six month study period will be excluded.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Omega 3 | 6 months
  Aim: To demonstrate the short-term multi focal electroretinogram (mfERG) effect of oral omega-3-fatty acids in the triglyceride form on dry age-related macular degeneration (AMD).
  Null hypothesis: Omega-3-fatty acids do not affect the mfERGs of patients with dry AMD.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Ho, MD, Principal Investigator — Retina Specialist
Locations (1):
- Mid Atlantic Retina, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gerstenblith AT, Baskin DE, Shah CP, Wolfe JD, Fineman MS, Kaiser RS, Ho AC. Electroretinographic effects of omega-3 Fatty Acid supplementation on dry age-related macular degeneration. JAMA Ophthalmol. 2013 Mar;131(3):365-9. doi: 10.1001/jamaophthalmol.2013.642. PMID 23494041